CLINICAL TRIAL: NCT01669837
Title: Cyanoacrylate Fixation for Laparoscopic Repair of Inguinal Hernias: a Prospective, Multicenter Registry
Brief Title: An Efficiency/Safety Study of Surgical Tissue Glue to Treat Inguinal Hernias
Status: Completed | Type: Observational
Sponsor: Duomed (Industry)
Responsible Party: Sponsor
Other Study IDs: BM-IFA-06
Record Dates: First submitted 2012-08-17; First posted 2012-08-21 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Inguinal Hernia
Keywords: Inguinal hernia; Laparoscopy; Surgical tissue glue
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient group: Administration of surgical tissue glue.
  Interventions: Device: Mesh fixation with surgical tissue glue

INTERVENTIONS:
Device: Mesh fixation with surgical tissue glue — Laparoscopic inguinal hernia repair using surgical tissue glue for mesh fixation

SUMMARY:
Prospective, multicenter, observational registry to collect data of laparoscopic inguinal hernia repair using surgical tissue glue fixation. The objective is to determine the prevalence of chronic pain at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patient is older than 18 years.
* Written informed consent is obtained from patient.
* Patient is able to complete the EQ-5D questionnaire.
* Patient has a primary unilateral or primary bilateral inguinal hernia- Mesh fixation is established with solely surgical tissue glue (Ifbond™).

Exclusion Criteria:

* Patient has a recurrent inguinal hernia.
* Patient is treated using the Lichtenstein technique.
* Mesh fixation with sutures, tacks, absorbable tacks or clips.
* Patient is allergic to components of surgical tissue glue (Ifbond™).
* Patient has a life expectancy of less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a primary inguinal hernia
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | up to 1 year
  Prevalence of postoperative pain evaluated by patient self-assessment using a visual analog scale.

SECONDARY OUTCOMES:
Intraoperative complications | 1 day
  Complications such as bowel injury, major bleeding, complications due to anesthesia, nerve damage, lesion of vas deferens.
Postoperative complications | Up to 30 days after index-procedure
  Local numbness, hematoma, seroma, wound infection, mesh infection, hernia recurrence.
Analgesic intake | Discharge, 5 weeks
  Intake of analgesics.
Quality of life (QOL) | Preoperative, 5 weeks, 1 year
  QOL assessed by EQ-5D questionnaire.
Freedom from hernia-related reinterventions | 1 year
  Reinterventions at 1 year after index-procedure assessed by means of a questionnaire.
Late complications | 1 year
  Local numbness, groin discomfort, hernia recurrence, sexual dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Van der Speeten, MD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium